CLINICAL TRIAL: NCT03338647
Title: Randomized Study of Stereotactic Body Radiation Therapy (SBRT) Versus Transarterial Chemoembolization (TACE) in Hepatocellular Carcinoma
Brief Title: SBRT or TACE for Advanced HCC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Aarhus (Other)
Collaborators: International Atomic Energy Agency (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UAarhus HCC
Record Dates: First submitted 2017-11-01; First posted 2017-11-09 (Actual); Last update posted 2021-12-02 (Actual); Status verified 2021-05

CONDITIONS: Hepatocellular Carcinoma
Keywords: Stereotactic body radiation therapy; transarterial chemoembolization; SBRT; TACE
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TACE (Active Comparator): Transarterial chemoembolization with drug eluted beads or doxorubicin/lipiodol
  Interventions: Drug: DEB
- SBRT (Experimental): Stereotactic radiation therapy with risk adapted dose prescription
  Interventions: Radiation: SBRT

INTERVENTIONS:
Drug: DEB — Infusion of DEB or doxorubin/lipiodol through catheter in the hepatic artery
  Other Names: doxorubicin
  Arms: TACE
Radiation: SBRT — High precision radiation therapy to the liver tumor(s)
  Arms: SBRT

SUMMARY:
Randomized study of stereotactic body radiation therapy (SBRT) versus transarterial chemoembolization (TACE) in locally advanced hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* HCC (biopsy or radiological diagnostic (>1 cm, enhancing in arterial phase and wash-out in later phases).
* Number of lesions: not more than 3 lesions
* Lesion size: up to 10 cm for a single lesion (and up to 10 cm cumulative diameter, if there is more than 1 lesion)
* Child-Pugh A or B (<7) on examination within 6 weeks prior to study entry
* BCLC Stage A/B
* Must be fit (eligible) for SBRT and TACE
* Unsuitable/unwilling for resection or transplant or radiofrequency ablation (RFA) or if these options are not available
* Distance between GTV (lesion) and luminal structures (including esophagus, stomach, duodenum, small or large bowel) is >10 mm
* All blood work obtained within 2 weeks prior to study entry with adequate organ function defined as follows:

  * Absolute neutrophil count (ANC) ≥ 1,500 cells/mm3
  * Platelets ≥50,000 cells/mm3
  * Hemoglobin ≥ 8.0 g/dl (Note: The use of transfusion or other intervention to achieve Hgb ≥ 8.0 g/dl is acceptable.)
  * Total bilirubin < 2 mg/dL
  * Prothrombin time/INR < 1.4 (unless on Coumadin/Warfarin)
  * Albumin ≥ 28 g/L
  * AST (and ALT) < 5 times ULN
  * Serum creatinine ≤ ULN or creatinine clearance ≥ 60 mL/min
  * Left-ventricular ejection fraction >50% (cardiac ejection fraction should be measured in case of history of cardio-vascular disease.
  * May have had previous surgery, ethanol injection and RFA to the liver

Exclusion Criteria:

* • Not suitable for clinical trial or follow-up

  * Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 2 years (Note that carcinoma in situ of the breast, oral cavity, or cervix are all permissible). No active cancer therapy.
  * Unsuitable for or refractory to transarterial hepatic chemo-embolization (TACE)

    * Non-enhancing HCC on CT or CT-angio or
    * Portal vein thrombosis/macroscopic venous invasion
  * Arterio-portal and arterio-venous fistulas observed on pre-study imaging (if it is found during the TACE, the fistula may be embolized before injection of the drug).
  * Evidence of metastatic disease including nodal or distant metastases.
  * Previous TACE or radiation to the liver (including SIRT)
  * Life-threatening condition (including untreated HIV and active hepatitis B/C)

    * Detectable HBeAg and HBV viral load > 20,000 IU/mL or
    * HBeAg-negative chronic hepatitis B and HBV viral load >2,000 IU/mL
    * If HBV-DNA copy is higher than 500 copies/ml, anti-viral therapy, such as Entecavir followed by observation for 2 weeks.
    * If anti-HCV antibody is positive (may be false positive) and increased HCV viral load indicating active disease. Active HCV should be treated sufficiently before inclusion in the study. Below 2 million copies per milliliter (mL) is related to chronic hepatitis C that does not need antiviral therapy.
    * Patients with active hepatitis B or C should be on treatment for at least 4 weeks before inclusion in the trial
  * On sorafenib or other antineoplastic drug therapy within 7 days before inclusion (not accepted until time of progression).
  * Pregnancy or women of childbearing potential require a negative pregnancy test within 28 days

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2017-10-26 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression (total of local, intra- and extrahepatic) | 1 year
  Modified RECIST

SECONDARY OUTCOMES:
Response | 3 months
  Modified RESIST
Local control of treated tumor | 1 year
  Modified RECIST
Intrahepatic failure | 1 year
  Intrahepatic failure (more than 1 cm away)
Extrahepatic failure | 1 year
  Modified RECIST
Overall survival | 1 year
  Overall survival
Treatment related toxicity | 1 year
  Tox CTC Ver 4.0
Cost-benefit | 1 year
  $ spend on hospitalization and treatment of complications after the treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Medanta, Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Yes
Upon request
Supporting Information: Study Protocol